CLINICAL TRIAL: NCT02314273
Title: Effect of Treatment Using rhIL-11 in Patients With Thrombocytopenia After Chemotherapy for Childhood Acute Lymphoblastic Leukemia
Brief Title: Effect of rhIL-11 in Patients With Thrombocytopenia for Childhood ALL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBK-10-01
Record Dates: First submitted 2014-07-25; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Pancytopenia Due to Chemotherapy
MeSH Terms: interventions — oprelvekin; Interleukin-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhIL-11 group (Experimental): patients receive rhIL-11(50 mcg/kg，subcutaneously)after standard chemotherapy，once a day for 10 days or until platelet count ≥80,000/mL
  Interventions: Drug: rhIL-11
- control group (No Intervention): control group

INTERVENTIONS:
Drug: rhIL-11 — patients receive rhIL-11(50 mcg/kg，subcutaneously)after standard chemotherapy，once a day for 10 days or until platelet count ≥80000/mL
  Other Names: Recombinant Human Interleukin-11
  Arms: rhIL-11 group

SUMMARY:
The goal of this clinical research study is to find out if rhIL-11（Interleukin 11） may increase the platelet count in Childhood patients with acute lymphocytic leukemia (ALL) who develop low platelet counts while receiving standard CAT（cyclophosphamide+Cytosine arabinoside+mercaptopurine，7d） therapy.

DETAILED DESCRIPTION:
Group A：patients receive rhIL-11(50 mcg/kg，subcutaneously)after standard chemotherapy，once a day for 10 days or until platelet count ≥80,000/mL Group B：control group

ELIGIBILITY:
Inclusion Criteria:

* new diagnosis of ALL
* TBIL≤34umol/L，Cr≤120umol/L，a normal EF
* age <18 years

Exclusion Criteria:

* patients with uncontrolled infection
* patients with Acute congestive heart failure or chronicity cardiorespiratory functional defect or serious cardiac arrhythmias

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
platelet infusion | 14 days
  frequency of platelet infusion

SECONDARY OUTCOMES:
hemorrhagic tendency | 14 days
  conditions of bleeding
infection | 14 days
  incident of infection during 14d after chemotherapy
remission rate | 14 days
  remission rate during 14d after chemotherapy
platelet Count | 14 days
  recovery of peripheral platelet count

CONTACTS AND LOCATIONS:
Overall Officials: Tang Jingyan, M.D., Study Chair — Shanghai Children's Medical Center
Locations (5):
- China (5):
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Soochow University Affiliated Children's Hospital, Suzhou, Jiangsu
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality